CLINICAL TRIAL: NCT05664035
Title: Detection of Specific Polysaccharide Antibody Deficiency in Adult Patients With Unexplained Recurrent and/or Severe Bacterial Infections
Brief Title: SPAD in Adult Patients
Acronym: DETECT
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: French Healthcare network for rare immune and hematological disorders (MARIH) (Unknown); Takeda (Industry); VitalAire (Industry); Laboratoire français de Fractionnement et de Biotechnologies (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021_0699; 2022-A00574-39 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2022-12-15; First posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Specific Antibody Deficiency; Predominantly Antibody Deficiencies
Keywords: Specific Antibody Deficiency; Predominant antibody deficiencies; Ig replacement therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Case group: 18 to 65 year old patients with a history of recurrent bacterial infections of upper and/or lower respiratory tract for at least 2 years
  Interventions: Biological: Diagnosis of SPAD using immunization with PPV23

INTERVENTIONS:
Biological: Diagnosis of SPAD using immunization with PPV23 — Diagnosis of SPAD using immunization with PPV23

SUMMARY:
The DETECT study aims to demonstrate the importance of detecting SPAD in adult patients with recurrent benign and/or severe unexplained bacterial upper/lower respiratory tract infections. Unlike children in whom the deficit may be transient, long-term strategies are warranted in SPAD adult patients to prevent severe infections and lung disability. Beyond the diagnosis of this still unrecognized PID in adult patients, we want to assess the impact of prophylactic antibiotics or IgRT on infections prevention and on quality of life in adult patients with the most severe clinical phenotypes, recurrent infections with high frequency of antibiotics take and/or recurrent infections with complications like bronchiectasis and/or severe infections requiring hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 year old patients
* With a history of recurrent bacterial infections of upper and/or lower respiratory tract for at least 2 years, and fulfilling the specific following criteria:
* Recurrent benign infections currently requiring 6 courses of antibiotics /year or more, or Bilateral bronchiectasis/bronchiolitis (after exclusion of cystic fibrosis and ciliary dyskinesia) AND recurrent benign infections currently requiring 3 courses of antibiotics /year or more or A history of severe upper/lower respiratory tract bacterial infection, and/or invasive infection with Streptococcus pneumonia, Streptococcus pyogenes or Haemophilus influenzae, which required hospitalization in the last 2 years, AND recurrent benign infections currently requiring 3 courses of antibiotics /year.
* Normal serum IgG, IgA, IgM and IgG subclasses levels, normal CH50 and serum complement C3 and C4 proteins levels, normal T cells count
* Normal B cell count, normal serum protein electrophoresis and immunofixation. (* excepted for Pseudomonas aeruginosa colonization)

Exclusion Criteria:

* Any general condition that predisposes to infections: solid or hematological malignancies, diabetes mellitus, severe alcohol or intravenous drug abuse, chronic liver or kidney failure, human immunodeficiency virus infection, anatomic or functional asplenia, drug-induced 1 neutropenia, or solid organ or hematopoietic stem cell transplantation;
* Any local predisposing factor to infections: cigarette smoking (> 10 pack-year and/or 5 cigarettes/day), underlying infection (tuberculosis, influenza…), chronic obstructive pulmonary disease, oral, dental or skin conditions favorizing infections, streptococcal skin infections
* Any other SID or PID diagnosed before inclusion
* Pregnancy
* PPV23 administration in the last 2 years (risk of hyporesponsiveness)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen in Pneumology, Immunology, ENT or Infectious Diseases departments
Sampling Method: Non-Probability Sample
Enrollment: 99 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of SPAD according to the AAAAI proposed consensus criteria for an impaired selective response to PS using immunization with PPV23 and assessment of anti-PnPS IgG response by the serotype-specific WHO-standardized ELISA 4 | to 8 weeks after immunization

SECONDARY OUTCOMES:
frequency of associated autoimmune or allergic diseases. | Througth study completion, an average 24 months
number of courses of antibiotics in the 12 months following IgRT start compared to the 12 months before IgRT | Througth study completion, an average 24 months
SF-36 questionnaire, number of missed work or school/university days in the 12 months following IgRT start compared to the 12 months before IgRT | Througth study completion, an average 24 months
frequency of courses of antibiotics in the 6 months following prophylaxis start compared to the 12 months before and/or number of patients switched to IgRT during the first 12 months. | Througth study completion, an average 24 months
SF-36 questionnaire, number of missed work or school/university days in the 12 months following prophylaxis start (or at the end of prophylactic antibiotics) compared to the 12 months before | Througth study completion, an average 24 months
Biological collection | Througth study completion, an average 24 months
  To collect serum and mononuclear cells for future research projects in SPAD and undiagnosed patients

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume LEFEVRE, MD,PhD, Principal Investigator — University Hospital, Lille